CLINICAL TRIAL: NCT01062178
Title: The Comparison of Accuracy of Contrast Enhanced Ultrasound on Diagnosis of Small Renal Masses and Distinguishing Renal Cell Carcinomas From Other Renal Masses, With Biopsy
Brief Title: Efficacy of Ultrasound Contrast Agent to Assess Renal Masses
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Lantheus Medical Imaging (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 08-0512-CE
Record Dates: First submitted 2010-01-22; First posted 2010-02-04 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-03

CONDITIONS: Renal Cell Carcinoma
Keywords: Small renal Mass; Contrast Enhanced Ultrasound; Renal Cell Carcinoma; noninvasive diagnosis of RCC
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — perflutren

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- comparison to biopsy (Experimental): Comparing contrast enhanced US with biopsy result
  Interventions: Drug: Definity

INTERVENTIONS:
Drug: Definity — Definity is the contrast agent which is going to be injected in a bolus and infusion forms during the ultrasound performance.

SUMMARY:
Patients with an incidentally discovered small renal masses (SRM) < 4 cm in diameter are included. All patients will undergo biopsy for tissue diagnosis. Most patients will be followed by imaging. Study intervention includes low MI US to be performed following both bolus and infusion injection of Definity contrast. Presence and absence of vascularity, pattern of vascularity, and TIC values will be correlated with the final pathology to find features differentiating benign from malignant masses.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed Renal mass < 4 cmm, who are going to undergo diagnostic CT, MRI or biopsy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2009-10; Primary Completion 2012-10 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
biopsy | 12 to 18 months

CONTACTS AND LOCATIONS:
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No